CLINICAL TRIAL: NCT06619327
Title: Resilient Together for Dementia: a Live Video Resiliency Dyadic Intervention for Persons with Dementia and Their Care-partners Early After Diagnosis
Brief Title: Resilient Together for Dementia (RT-D)
Acronym: RT-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sarah Bannon, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 23-0519-0001; 1K23AG075188 (NIH)
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Dementia
Keywords: Dementia; Care partners; Dyads; Emotional distress; Quality of life; Couples
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Resilient Together for Dementia (Experimental): The research team will compare two programs to reduce emotional distress among couples after dementia diagnosis.
  Interventions: Behavioral: Resilient Together for Dementia; Behavioral: MEUC

INTERVENTIONS:
Behavioral: Resilient Together for Dementia — RT-D has been developed based on feedback from couples and dementia clinicians as well as prior successful dyadic interventions. RT-D was developed based on the Recovering Together (RT) dyadic intervention for acute neurological illnesses and is being adapted to address the needs of couples navigating new dementia diagnoses.
  Other Names: RT-D
Behavioral: MEUC — The MEUC condition was also developed based on the comparison trial in the Recovering Together dyadic intervention, and was adapted based on feedback from prior studies. The program is self-guided and provides educational information similar to the RT-D condition, but with no skills practice or weekly sessions with a therapist.
  Other Names: Minimally enhanced usual care

SUMMARY:
This study will evaluate the feasibility and preliminary efficacy of the novel Resilient Together for Dementia (RT-D) intervention for couples following dementia diagnoses. The primary target is emotional distress, and the program aims to prevent chronic distress in at-risk couples.

DETAILED DESCRIPTION:
Both persons living with dementia and their spousal care-partners experience high levels of clinically elevated emotional distress, which can become chronic without treatment and negatively impact the health, quality of life, communication, and care-planning of both partners. A tailored dyadic intervention, such as the proposed Resilient Together for Dementia, delivered over live video to this at risk population has the potential to prevent chronic emotional distress and preserve quality of life for PWDs and their loved ones.

A pilot feasibility randomized control trial (RCT; Aim 3; NIA Stage 1B; N=50 dyads) will be conducted of the refined RT-D versus a minimally enhanced educational control (MEUC, educational pamphlet). Primary outcomes will be feasibility, credibility, and acceptability markers to inform a hybrid efficacy effectiveness R01 (year 4) of RT-D vs. MEUC (NIA Stage II). In this subsequent R01, the researcher will examine RT-D's impact on emotional distress and quality of life outcomes and test mechanisms of change (individual and interpersonal resiliency skills) through mediation and moderation. The researcher will revise the approach if feasibility benchmarks are not met.

ELIGIBILITY:
Inclusion Criteria:

* Recent (~3 month) chart documented ADRD diagnosis,
* ADRD symptom onset after age 65
* Cognitive assessment scores and symptoms consistent with early stage dementia, as determined by the Clinical Dementia Rating Scale scores of .5 or 1.0
* Cognitive awareness of their problems (as determined by the treating neurologist), and ability to understand study and research protocol, as determined by a standardized teach-back method assessment

Additional inclusion criteria for dyads are:

* English speaking adults (18 years or older)
* Dyad lives together
* At least one partner endorses clinically significant emotional distress during screening (>7 on Hospital Anxiety and Depression scale subscales or <5 on the Geriatric Depression Scale)

Exclusion Criteria:

* Patient is deemed inappropriate by the neurology team
* Either partner has a co-occurring terminal illness
* Patient was diagnosed with forms of dementia with clinical profiles that would preclude participation (e.g., Frontotemporal Dementia- behavioral variant), as determined by treatment team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants screened | After each dyad completion, throughout study of 6-8 weeks
  Feasibility of recruitment - recruitment will be monitored by screening clinic visits for potentially eligible individuals and review recruitment progress in weekly meetings to promote completion within the study time frame. The research team will measure with the proportion of participants screened.
Proportion of participants who consent or not consent to participate | After each dyad completion, throughout study of 6-8 weeks
  Feasibility of consent - by keeping a record of all individuals who complete screening that consent, refuse to consent, and the reasons for refusal will be monitored and will review progress in weekly team meetings. The research team will measure with the proportion of participants who consent or not consent to participate
Proportion of sessions participants attend | After each dyad completion, throughout study of 6-8 weeks
  The number of sessions that enrolled dyads attend as well as missed sessions, treatment dropouts, and reasons for nonattendance will be monitored and will review progress in weekly meetings. The research team will measure with the proportion of sessions participants attend.
Credibility and Expectancy Questionnaire (CEQ) | After each dyad completion, throughout study of 6-8 weeks
  A scale measuring treatment expectancy and rationale credibility for use in clinical outcome studies. Full scale from 0-10, with higher score indicating higher treatment expectancy
Client Satisfaction Questionnaire | After each dyad completion, throughout study of 6-8 weeks
  A 3-item questionnaire assessing participants' satisfaction with participation in the study. Full scale from 0-12, with higher score indicating greater satisfaction.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | Baseline to posttest (6-8 weeks)
  A 14-items scale with responses scored from 0-3, scores for each subscale from 0 (normal) to 21 (severe symptoms). Full scale score is 0 to 42, with higher score indicating more emotional distress.
Geriatric Depression Scale | Baseline to posttest (6-8 weeks)
  A 15-item scale with yes/no responses, total scores range from 0 to 15. Scores of 0-4 are considered normal, 5-8 indicate mild depression, 9-11 suggest moderate depression, and 12-15 indicate severe depression. Higher scores indicate more severe depressive symptoms.
Perceived Stress Scale | Baseline to posttest (6-8 weeks)
  A 10-item questionnaire, each item scored 0 (never) to 4 (very often), full scale from 0-40, with higher score indicating higher perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Bannon, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Brain Injury Research Center at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact sarah.bannon@mountsinai.org